CLINICAL TRIAL: NCT01639235
Title: Cardiopulmonary Effects of Secondhand Smoke Exposure on Flight Attendants
Brief Title: Effects of Secondhand Smoke on Flight Attendant Health
Acronym: FAMRI
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Flight Attendant Medical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 14-13934; FAMRI (Other Grant/Funding Number: FAMRI (Flight Attendant Medical Research Institute)); 146312 (Other: University of California, San Francisco)
Record Dates: First submitted 2012-07-09; First posted 2012-07-12 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Cardiopulmonary Disease
Keywords: Secondhand Smoke; Flight Attendants; Lung function; Cardiac function; Reproductive health
MeSH Terms: conditions — Pulmonary Heart Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — There is an optional blood draw blood portion to the research study. A sample is collected from the interested flight attendant. The majority of the sample is processed and stored in the FAMRI biorepository for future research purposes to identify biomarkers of cardiovascular risk and secondhand smoke. The remainder of the sample is analyzed for the flight attendant. A lipid profile is sent to the flight attendant participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a study on a population of flight attendants who were exposed to occupational secondhand tobacco smoke (SHS). This research will examine associations between flight attendant SHS exposure and development of respiratory illnesses, reproductive problems, and cardiovascular diseases.

DETAILED DESCRIPTION:
The main hypothesis of this study is that exposure to the secondhand tobacco smoke (SHS) in the confined workspace of commercial aircraft prior to the ban of cigarette smoking is responsible for long-term damage on the health of nonsmoking flight attendants. We will compare the data collected from our pre-ban flight attendant participants to age-matched, nonsmoking controls from the NHANES (National Health and Nutrition Examination Survey) database. The results of our study should permit us to determine if SHS exposure is the cause of long-term increased cardiovascular morbidity and risk, as well as increased susceptibility to respiratory illnesses.

ELIGIBILITY:
Inclusion Criteria:

1. Never smoker flight attendants who began working for airlines before the smoking ban on aircrafts went into effect. Never smoker is defined as those with history of tobacco use of less than 100 cigarettes in their lifetime.
2. SHS exposure for at least 1 year while working with the airlines.

Exclusion Criteria:

1. Less than 1 year of occupational exposure to SHS
2. Smoking more than 100 cigarettes over a lifetime

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a cross-sectional observational study of flight attendants exposed to secondhand tobacco smoke.
Sampling Method: Non-Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2005-01-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Characterize the long-term effects of SHS on lung and cardiovascular function in pre-ban flight attendants | 25 minutes
  A spirometry test is performed by the Clinical Research Coordinator to establish the lung function of the flight attendant participant and medical assistants from the cardiovascular care clinic administer a 12-lead non-invasive electrocardiogram.

SECONDARY OUTCOMES:
Clinical Examination | 30 min
  The cardiologist performs a noninvasive assessment of the patient's vascular function, which includes a brief physical examination, blood pressure measurement, pulse, and oxygen level.
Characterize the long term effects of prolonged flight time and SHS on reproductive health | 10 minutes
  Flight attendants fill out the electronic Exposure Questionnaire prior to their appointments. Part of the Questionnaire is a section on reproductive health. The answers to these survey questions in addition to information gathered and saved in the local medical record system (APeX) during the clinic visit are used for analysis on reproductive health of flight attendants.
Characterize the biomarkers of SHS exposure | 10 minutes
  A 45 mL blood specimen is drawn from interested patients to be stored in the research lab as well as analyzed in a University of California, San Francisco (UCSF) laboratory. Results of the blood analysis performed in the research labs, such as secondhand smoke biomarkers and advanced lipid biomarkers, will not be shared with the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Redberg, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No